CLINICAL TRIAL: NCT00080808
Title: A Randomized Phase II Trial Evaluating the Importance of Early Erectile Dysfunction Rehabilitation and Unilateral Autologous Sural Nerve Sparing Radical Prostatectomy Clinically Localized Prostate Cancer
Brief Title: Nerve-Sparing Radical Prostatectomy With or Without Nerve Grafting Followed by Standard Therapy for Erectile Dysfunction in Treating Patients With Localized Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: ID01-304; P50CA090270 (NIH); P30CA016672 (NIH); MDA-ID-01304 (Other: UT MD Anderson Cancer Center); CDR0000355366 (Registry Identifier: NCI PDQ)
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Last update posted 2012-07-30 (Estimated); Status verified 2012-07

CONDITIONS: Prostate Cancer
Keywords: perioperative/postoperative complications; sexual dysfunction and infertility; sexuality and reproductive issues; adenocarcinoma of the prostate; stage I prostate cancer; stage II prostate cancer; prostaglandin E1; papaverine; phentolamine; Nerve-sparing radical prostatectomy; nerve grafting
MeSH Terms: conditions — Prostatic Neoplasms; Postoperative Complications; Sexual Dysfunction, Physiological; Infertility; Sexuality | interventions — Alprostadil; methyl N-acetylsibirosaminide; Papaverine; Phentolamine; Sildenafil Citrate; Prostatectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm I (Active Comparator): Patients undergo unilateral cavernous nerve-sparing radical prostatectomy with unilateral autologous interposition sural nerve grafting.
  Interventions: Drug: Alprostadil (E1); Drug: Papaverine; Drug: Phentolamine mesylate; Drug: Sildenafil citrate; Procedure: conventional surgery
- Arm II (No sural nerve grafting) (Active Comparator): Patients undergo unilateral cavernous nerve-sparing radical prostatectomy (without sural nerve grafting) and erectile dysfunction rehabilitation as in arm I.
  Interventions: Drug: Alprostadil (E1); Drug: Papaverine; Drug: Phentolamine mesylate; Drug: Sildenafil citrate; Procedure: conventional surgery

INTERVENTIONS:
Drug: Alprostadil (E1) — Beginning 6 weeks after surgery, intracavernous Triplemix (prostaglandin E1, papaverine, and phentolamine) injected twice weekly
  Other Names: Prostaglandin E1; PGE1
Drug: Papaverine — Beginning 6 weeks after surgery, intracavernous Triplemix (prostaglandin E1, papaverine, and phentolamine) injected twice weekly
  Other Names: Paverine Injection; Papaverine Hydrochloride Injection
Drug: Phentolamine mesylate — Beginning 6 weeks after surgery, intracavernous Triplemix (prostaglandin E1, papaverine, and phentolamine) injected twice weekly
Drug: Sildenafil citrate — Oral sildenafil as needed
  Other Names: Viagra
Procedure: conventional surgery — Unilateral cavernous nerve sparing radical retropubic prostatectomy
  Other Names: prostatectomy

SUMMARY:
RATIONALE: Nerve-sparing radical prostatectomy with nerve grafting followed by standard therapies for erectile dysfunction may be effective in helping patients with prostate cancer improve sexual satisfaction and quality of life. It is not yet known whether erectile dysfunction therapy and nerve-sparing prostatectomy are more effective with or without nerve grafting.

PURPOSE: This randomized phase II trial is studying nerve grafting and standard therapy to see how well they work compared to standard therapy alone in treating erectile dysfunction in patients undergoing nerve-sparing radical prostatectomy for localized prostate cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare the efficacy of erectile dysfunction rehabilitation and unilateral cavernous nerve-sparing radical prostatectomy with versus without unilateral autologous interposition sural nerve grafting in patients with clinically localized prostate cancer.
* Compare potency rates in patients treated with these regimens.
* Compare erection quality in patients treated with these regimens.
* Compare time to return of spontaneous erectile activity in patients treated with these regimens.
* Compare the feasibility of these regimens in these patients.
* Compare quality of life and sexual satisfaction in patients treated with these regimens.
* Compare changes in penile erectile length and circumference in patients treated with these regimens.
* Compare the relative morbidity of patients treated with these regimens.

OUTLINE: This is a randomized, open-label study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients undergo unilateral cavernous nerve-sparing radical prostatectomy with unilateral autologous interposition sural nerve grafting.

Beginning 6 weeks after surgery, patients undergo erectile dysfunction rehabilitation comprising any of the following: oral sildenafil (as occasion requires), use of vacuum erection device over 10 minutes once daily, intracavernous Triplemix (prostaglandin E1, papaverine, and phentolamine) injected twice weekly, or MUSE (suppository in urethra for erections) therapy. Erectile dysfunction rehabilitation may continue for up to 2 years or until return of adequate spontaneous erectile activity.

* Arm II: Patients undergo unilateral cavernous nerve-sparing radical prostatectomy (without sural nerve grafting) and erectile dysfunction rehabilitation as in arm I.

In both arms, treatment continues in the absence of unacceptable toxicity.

Quality of life and sexual history are assessed at baseline, at 6 weeks postoperatively, at 4, 8, 12, and 16 months, and then every 4 months for 2 years or until return of spontaneous erectile activity.

Patients are followed every 4 months for 2 years.

PROJECTED ACCRUAL: A total of 200 patients (120 for arm I and 80 for arm II) will be accrued for this study.

ELIGIBILITY:
Inclusion Criteria:

1. Patient must be a candidate for a unilateral nerve sparing radical retropubic prostatectomy. a) Gleason score 7 or less in the cores on the side to be spared
2. Patient must have no discernable preoperative erectile dysfunction, defined as the ability to have successful penetration on at least 75% of attempts.
3. Patient must be </= 65 years of age at the time of study enrollment.
4. Patient must have no peripheral neuropathy precluding procurement of a sural nerve graft
5. Patient must have no significant psychiatric illness or demonstrable vasculogenic source of impotence.
6. No prior history of pelvic irradiation or androgen deprivation therapy (LHRH agonists or anti-androgens)

Exclusion Criteria:

Max Age: 65 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2001-08; Primary Completion 2006-07 (Actual); Study Completion 2009-07 (Actual)

PRIMARY OUTCOMES:
Potency rate at 2 years after surgery | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Christopher G. Wood, MD, Study Chair — M.D. Anderson Cancer Center
Locations (1):
- M.D. Anderson Cancer Center at University of Texas, Houston, Texas, United States

REFERENCES:
- [Result] Davis JW, Chang DW, Chevray P, Wang R, Shen Y, Wen S, Pettaway CA, Pisters LL, Swanson DA, Madsen LT, Huber N, Troncoso P, Babaian RJ, Wood CG. Randomized phase II trial evaluation of erectile function after attempted unilateral cavernous nerve-sparing retropubic radical prostatectomy with versus without unilateral sural nerve grafting for clinically localized prostate cancer. Eur Urol. 2009 May;55(5):1135-43. doi: 10.1016/j.eururo.2008.08.051. Epub 2008 Sep 2. PMID 18783876
- See also: UT MD Anderson Cancer Center Website — http://www.mdanderson.org